CLINICAL TRIAL: NCT05121766
Title: Feasibility Pilot Clinical Trial of Omega-3 (EPA+DHA) Supplement vs. Placebo for Post-Acute Sequelae of Coronavirus-19 (COVID-19) Recovery Among Health Care Workers
Brief Title: Feasibility Pilot Clinical Trial of Omega-3 Supplement vs. Placebo for Post Covid-19 Recovery Among Health Care Workers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Challenges in enrollment
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2020-1166
Record Dates: First submitted 2021-11-15; First posted 2021-11-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: post-acute sequelae of covid-19; post- covid syndrome; long covid syndrome; healthcare workers; post-covid symptoms; quality of life; omega-3
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Docosahexaenoic Acids; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Everybody but the pharmacy team dispensing the drug will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study arm - Omega 3 supplement (Experimental): Omega-3 (EPA+DHA) - Dose is 2,100mg per day via 3 mini-capsules, 2x/day (a total of 6 mini-capsules per day). Each capsule has 252mg of EPA and 102mg of DHA.
  Interventions: Drug: Omega-3 (EPA+DHA)
- Control arm - placebo (Placebo Comparator): 3 Soybean Oil Placebo capsules 2x/day (a total of 6 mini-capsules per day).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3 (EPA+DHA) — Dose is 2,100mg per day via 3 mini-capsules, 2x/day (a total of 6 mini-capsules per day).
  Each capsule has 252mg of EPA and 102mg of DHA.
  Other Names: fish oil
  Arms: Study arm - Omega 3 supplement
Drug: Placebo — 3 Soybean Oil Placebo capsules
  Arms: Control arm - placebo

SUMMARY:
This is a two-arm, double blind randomized 12-week study to supplement omega-3 (Eicosapentaenoic acid - EPA + docosahexaenoic acid - DHA) among 100 adults (age 18+) who had coronavirus-19 (covid-19) and are experiencing possible after-effects from post-acute sequelae of covid-19 (also called post-covid syndrome or long covid syndrome).

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled trial (RCT) with two treatment arms:

Arm 1 - Omega-3 (Eicosapentaenoic acid - EPA + docosahexaenoic acid - DHA) - Dose is 2,100mg per day via 3 mini-capsules, 2x/day (a total of 6 mini-capsules per day). Each capsule has 252mg of EPA and 102mg of DHA.

Support for dosing:

* The American Heart Association (AHA) says taking up to 3 grams of fish oil daily in supplement form is considered safe;
* Up to 5,000mg of omega-3 fatty acids per day is considered safe;
* The U.S. Food and Drug Administration recommends consuming no more than 3 g/day of EPA and DHA combined, including up to 2 g/day from dietary supplements.

Arm 2 - Placebo - made from soybean oil (same dosing schedule as intervention arm)

ELIGIBILITY:
Inclusion Criteria:

* Team member at Hackensack Meridian Health
* Age: 18+
* Willing to provide informed consent
* Formal diagnosis of COVID-19 via Polymerase Chain Reaction (PCR)test (if home test was done, team member must confirm via PCR test)
* Outpatient treatment only for covid-19; no hospitalization (most team members will be vaccinated and may likely have milder case)
* Must be experiencing 1+ ongoing covid-19 symptom being measured in this study (respiratory symptoms (shortness of breath, cough), fatigue, loss of taste, loss of smell)
* Symptom(s) have persisted for more than 12 weeks after initial infection
* Symptom(s) coincided with covid-19 infection and were not present prior to covid-19 infection
* Does not have soy allergy
* Does not have allergy to fish
* Able to participate in bi-weekly surveys in Research Electronic Data Capture (REDCap)
* Able to take own blood pressure and record it in bi-weekly REDCap survey
* Willing to participate in 12-week study and be assigned to either intervention or placebo arm
* Not currently taking an omega-3 supplement or other high-dose supplement (over 2,000 IU) with potential for aiding recovery of long covid syndrome (e.g. zinc, Vit C, Elderberry).
* Able to take/swallow six mini-pills daily
* Able and willing to give a spot blood sample (2 drops) at baseline and end of study.

Exclusion Criteria:

* Not a Team Member at Hackensack Meridian Health
* Not age 18+
* Unwilling to provide informed consent/ declined to take part
* No formal diagnosis of COVID-19 via PCR test (if home test was done, team member must confirm via PCR test)
* Were hospitalized for treatment of covid-19
* Not experiencing 1+ ongoing covid-19 symptom being measured in this study (respiratory symptoms (shortness of breath, cough), fatigue, loss of taste, loss of smell)
* Symptom(s) have persisted for more than 12 weeks after initial infection
* Symptom(s) did not coincide with covid-19 infection and were present prior to covid-19 infection
* Does have soy allergy
* Does have allergy to fish
* Not able to participate in bi-weekly surveys in REDCap
* Able to take own blood pressure and record it in bi-weekly REDCap survey
* Not willing to participate in 12-week study and be assigned to either intervention or placebo arm
* Currently taking an omega-3 supplement or other high-dose supplement (over 2,000 IU) with potential for aiding recovery of long covid syndrome (e.g. zinc, Vit C, Elderberry).
* Unable to take/swallow six mini-pills daily
* Not able and not willing to give a spot blood sample (2 drops) at baseline and end of study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arunima Sarkar, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Susan Dara, Edison, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. BourBour F, Mirzaei Dahka S, Gholamalizadeh M, et al. Nutrients in prevention, treatment, and management of viral infections; special focus on Coronavirus [published online ahead of print, 2020 Jul 9]. Arch Physiol Biochem. 2020;1-10. doi:10.1080/13813455.2020.1791188 2. Ali N. Role of vitamin D in preventing of COVID-19 infection, progression and severity [published online ahead of print, 2020 Jun 20]. J Infect Public Health. 2020;S1876-0341(20)30531-1. doi:10.1016/j.jiph.2020.06.021 3. Colunga Biancatelli RML, Berrill M, Catravas JD, Marik PE. Quercetin and Vitamin C: An Experimental, Synergistic Therapy for the Prevention and Treatment of SARS-CoV-2 Related Disease (COVID-19). Front Immunol. 2020;11:1451. Published 2020 Jun 19. doi:10.3389/fimmu.2020.01451 4.Torjesen I. Covid-19: Public health agencies review whether vitamin D supplements could reduce risk. BMJ. 2020;369:m2475. Published 2020 Jun 19. doi:10.1136/bmj.m2475 5.Hribar CA, Cobbold PH, Church FC. Potential Role of Vitamin D in the Elderly to Resist COVID-19 and to Slow Progression of Parkinson's Disease. Brain Sci. 2020;10(5):284. Published 2020 May 8. doi:10.3390/brainsci10050284 6. NIH Workshop on Post-Acute Sequelae of COVID-19. Accessed 25 Jan 2021. Available at: https://www.niaid.nih.gov/news-events/workshop-post-acute-sequelae-covid-19 7. Mayo Clinic: COVID-19 (coronavirus): Long-term Effects. Accessed 8 Jan 2021 from https://www.mayoclinic.org/diseases-conditions/coronavirus/in-depth/coronavirus-long-term-effects/art-20490351 8. Jacobs LG, Gourna Paleoudis E, Lesky-Di Bari D, et al. Persistence of symptoms and quality of life at 35 days after hospitalization for COVID-19 infection. PLoS One. 2020;15(12):e0243882. Published 2020 Dec 11. doi:10.1371/journal.pone.0243882 9. Halpin SJ, McIvor C, Whyatt G, Adams A, Harvey O, McLean L, Walshaw C, Kemp S, Corrado J, Singh R, Collins T, O'Connor RJ, Sivan M. Postdischarge symptoms and rehabilitation needs in survivors of COVID-19 infection: A cross-sectional evaluation. J Med Virol. 2021 Feb;93(2):1013-1022. doi: 10.1002/jmv.26368. Epub 2020 Aug 17. PMID: 32729939. 10. Garrigues E, Janvier P, Kherabi Y, et al. Post-discharge persistent symptoms and health-related quality of life after hospitalization for COVID-19. J Infect. 2020;81(6):e4-e6. doi:10.1016/j.jinf.2020.08.029
- [Background] 11. CDC Morbidity and Mortality Weekly Report: Symptom Duration and Risk Factors for Delayed Return to Usual Health Among Outpatients with Covid-19 in a Multistate Health Care Systems Network - United States - March-June 2020. Accessed on 25 Jan 2021 from https://www.cdc.gov/mmwr/volumes/69/wr/mm6930e1.htm 12. Couzin-Frankel, J. From 'brain fog' to heart damage, COVID-19's lingering problems alarm scientists. July 31, 2020. Accessed 25 January 2021 from https://www.sciencemag.org/news/2020/07/brain-fog-heart-damage-covid-19-s-lingering-problems-alarm-scientists 13. Cooney, Elizabeth. Stat / Health Column: Long after the fire of a covid-19 infection, mental and neurological effects can still smolder. Accessed 26 Jan 2021 from https://www.statnews.com/2020/08/12/after-covid19-mental-neurological-effects-smolder/ 14. Puntmann VO, Carerj ML, Wieters I, et al. Outcomes of Cardiovascular Magnetic Resonance Imaging in Patients Recently Recovered From Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020;5(11):1265-1273. doi:10.1001/jamacardio.2020.3557 15. Carfì A, Bernabei R, Landi F, for the Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020;324(6):603-605. doi:10.1001/jama.2020.12603 16. Gemelli Against COVID-19 Post-Acute Care Study Group. Post-COVID-19 global health strategies: the need for an interdisciplinary approach. Aging Clin Exp Res. 2020 Aug;32(8):1613-1620. doi: 10.1007/s40520-020-01616-x. Epub 2020 Jun 11. PMID: 32529595; PMCID: PMC7287410. 17. Scaioli E, Liverani E, Belluzzi A. The Imbalance between n-6/n-3 Polyunsaturated Fatty Acids and Inflammatory Bowel Disease: A Comprehensive Review and Future Therapeutic Perspectives. Int. J. Mol. Sci. 2017; 18(12): e2619 18.Yaqoob, P. Mechanisms underlying the immunomodulatory effects of n-3 PUFA. Proc. Nutr. Soc. 2010; 69(3): 311-315 19.Rees D, Miles EA, Banerjee T, Wells SJ, Roynette CE, Wahle KW, Calder PC. Dose-related effects of eicosapentaenoic acid on innate immune function in healthy humans: A comparison of young and older men. Am. J. Clin. Nutr. 2006; 83: 331-342 20. Endres S, Ghorbani R, Kelley VE, Georgilis K, Lonnemann G, van der Meer JW, Cannon JG, Rogers TS, Klempner MS, Weber PC, Schaefer EJ, Wolff SM, Dinarello CA. The effect of dietary supplementation with n-3 polyunsaturated fatty acids on the synthesis of interleukin-1 and tumor necrosis factor by mononuclear cells. N. Engl. J. Med. 1989; 320: 265-271
- [Background] 21.Kelei Li, Tao Huang, Jusheng Zheng, Duo Li. Effect of Marine-Derived n-3 Polyunsaturated Fatty Acids on C-Reactive Protein, Interleukin 6 and Tumor Necrosis Factor a: A Meta-Analysis. PLOS ONE, 2014;9(2): e88103 22. Mogensen TH, Melchjorsen J, Hollsberg P, Paludan SR. Activation of NF-kappa B in virus-infected macrophages is dependent on mitochondrial oxidative stress and intracellular calcium: Downstream involvement of the kinases TGF-beta-activated kinase 1, mitogen-activated kinase/extracellular signal-regulated kinase kinase 1, and I kappa B kinase. J Immunol. 2003; 170(12): 6224- 6233 23.Beyazit Y, Purnak T, Kekilli M. Role of nitric oxide in the treatment of non-alcoholic fatty liver by omega-3 fatty acids. Aliment. Pharmacol. Ther. 2010; 32(2): 303-304 24. Adli M, Merkhofer E, Cogswell P, Baldwin AS. IKKalpha and IKKbeta each function to regulate NFkappaB activation in the TNF-induced/canonical pathway. PLoS One. 2010 Feb 25; 5(2): e9428 25. Sabater J, Masclans JR, Sacanell J, Chacon P, Sabin P, Plnas M. Effects of an omega-3 fatty acid enriched lipid emulsion on eicosanoid synthesis in acute respiratory distress syndrome (ARDS): A prospective, randomized, double-blind, parallel group study Nutr Metab (Lond). 2011; 8(1): 22. 26. Dushianthan A, Rebecca Cusack V, Burgess A, Grocott M, Calder P. Immunonutrition for Adults With ARDS: Results From a Cochrane Systematic Review and Meta-Analysis, Respiratory Care January 2020; 65(1): 99-110 27. Langlois P, D'Aragon F, Hardy G, Manzanares W. Omega-3 polyunsaturated fatty acids in critically ill patients with acute respiratory distress syndrome: A systematic review and meta-analysis. Nutrition. 2019; 61: 84-92 28. Chen H, Wang S, Zhao Y, Luo Y, Tong H, Su L. Correlation analysis of omega-3 fatty acids and mortality of sepsis and sepsis-induced ARDS in adults: data from previous randomized controlled trials. Nutr J. 2018; 17(1): 57 29. NBC News, NJ Gov. Murphy says state is hardest hit by coronavirus in U.S. May 12, 2020. Accessed at: https://www.nbcnews.com/video/new-jersey-gov-murphy-says-state-is-hardest-hit-by-coronavirus-in-u-s-83346501863 30. NJ Department of Health / Covid-19 Dashboard. Accessed 8 Jan 2021 from https://covid19.nj.gov/
- [Background] 31. Barrett, E.S., Horton, D.B., Roy, J. et al. Prevalence of SARS-CoV-2 infection in previously undiagnosed health care workers in New Jersey, at the onset of the U.S. COVID-19 pandemic. BMC Infect Dis 20, 853 (2020). https://doi.org/10.1186/s12879-020-05587-2 32. Gooch, Kelly. Becker's Hospital Review: Covid-19 Sidelines over 100 New Jersey Hospital Workers. Dec 2, 2020. Accessed on 27 Jan 2021 from https://www.beckershospitalreview.com/workforce/covid-19-sidelines-over-100-new-jersey-hospital-workers.html. 33. American Heart Association: Professional Heart Daily (13 March 2017. Omega-3 Polyunsaturated Fatty Acid (Fish Oil) Supplementation and the Prevention of Clinical Cardiovascular Disease. Available at: https://professional.heart.org/en/science-news/omega-3-polyunsaturated-fatty-acid-fish-oil-supplementation-and-the-prevention 34. Scientific Opinion on the Tolerable Upper Intake Level of eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA) and docosapentaenoic acid (DPA). (Source: EFSA Panel on Dietetic Products, Nutrition and Allergies (NDA) / 27 July 2012 https://doi.org/10.2903/j.efsa.2012.2815|) 35.U.S. Food and Drug Administration. Summary of qualified health claims subject to enforcement discretion. 2014. Available at: https://www.fda.gov/food/food-labeling-nutrition/qualified-health-claims-letters-enforcement-discretion 36. Insights From the OPERA Randomized Trial--Emmanuel Akintoye , Prince Sethi, William S. Harris , Paul A. Thompson , Roberto Marchioli , Luigi Tavazzi , Roberto Latini , Mias Pretorius , Nancy J. Brown , Peter Libby, Dariush Mozaffarian, Originally published5 Nov 2018https://doi.org/10.1161/CIRCOUTCOMES.118.004584Circulation: Cardiovascular Quality and Outcomes. 2018;11 37. n-3 Fatty acids affect haemostasis but do not increase the risk of bleeding: clinical observations and mechanistic insights: John K Wachira, Mark K Larson, William S Harris; PMID: 24472372, DOI: 10.1017/S000711451300425X 38. Elevated plasma glucose and lowered triglyceride levels from omega-3 fatty acid supplementation in type II diabetes ; K E Friday , M T Childs, C H Tsunehara, W Y Fujimoto, E L Bierman, J W Ensinck--Diabetes Care . 1989 Apr; 12(4):276-81. doi:10.2337/diacare.12.4.276. 39. Effects of Omega-3 Fatty Acid Supplementation on Glucose Control and Lipid Levels in Type 2 Diabetes: A Meta-Analysis, Cai Chen, 1 , 2 Xuefeng Yu, 1 and Shiying Shao 1 ,* Published online 2015 Oct 2. doi: 10.1371/journal.pone.0139565 40. Morris MC, Sacks F, Rosner B. Does fish oil lower blood pressure? A meta-analysis of controlled trials. Circulation. 1993;88(2):523-533. doi:10.1161/01.cir.88.2.523 41. Cleveland Heart Lab: Omega-3 Fatty Acids: A Natural Way to Lower Blood Pressure. Blog post 20 August 2015. Available at: https://www.clevelandheartlab.com/blog/horizons-omega-3-fatty-acids-a-natural-way-to-lower-blood-pressure/ 42. Overview of Omega-3 Fatty Acid Therapies; J. Chris Bradberry, PharmD and Daniel E. Hilleman, PharmD----PMID: 24391388 43. Link, R. Healthline blog: 8 Little-Known Side Effects of Too Much Fish Oil. 17 July 2018. Available at: https://www.healthline.com/nutrition/fish-oil-side-effects#section4 44. Khodarahmi M, Azadbakht L. Dietary fat intake and functional dyspepsia. Adv Biomed Res. 2016;5:76. Published 2016 Apr 21. doi:10.4103/2277-9175.180988

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm - Omega 3 Supplement: Omega-3 (EPA+DHA) - Dose is 2,100mg per day via 3 mini-capsules, 2x/day (a total of 6 mini-capsules per day). Each capsule has 252mg of EPA and 102mg of DHA.
  Omega-3 (EPA+DHA): Dose is 2,100mg per day via 3 mini-capsules, 2x/day (a total of 6 mini-capsules per day).
  Each capsule has 252mg of EPA and 102mg of DHA.
Period: Overall Study
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Started | 16 | 16
Completed | 8 | 10
Not Completed | 8 | 6
Not completed — Covid reinfection | 3 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients consented into the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] | 46.44 [27 to 62] | 47.25 [24 to 66] | 46.84 [24 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 14 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Study for Omega-3 Fatty Acid Supplementation v. Placebo in Adult Patients to Limit Long Covid Syndrome - Compliance as Captured by the Number of Participants Who Remain Compliant for the Whole Duration of the Study by Taking All Pills Daily
Description: Number of participants who remain compliant for 12 weeks
Time Frame: 12 weeks
Population: Number of participants who completed the 12-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Number analyzed (Participants) | 16 | 16
Participants | 8 | 10

2. Primary Outcome: Feasibility Study for Omega-3 Fatty Acid Supplementation v. Placebo in Adult Patients to Limit Long Covid Syndrome - Recruitment as Illustrated by the Number of Screen Failures (Potential Participants Approached But Not Interested in Participating).
Description: Number of participants who expressed interest in learning about the study
Time Frame: 6 months recruitment efforts (starting on actual study start date)
Population: Potential participants expressing interest in the study
Measure: Count of Participants; unit: Participants
Groups:
- Healthcare Workers Interested in Participating: Number of potential participants that were informed about the study
Arm/Group | Healthcare Workers Interested in Participating
Number analyzed (Participants) | 93
Participants
  Interested to participate but not eligible | 60
  Chose not to participate after learning more about the study | 1
  Signed consent | 32

3. Primary Outcome: Feasibility Study for Omega-3 Fatty Acid Supplementation v. Placebo in Adult Patients to Limit Long Covid Syndrome - Retention as Illustrated by the Number of Participants That Initiate But do Not Complete the Study.
Description: Number of participants who initiate but do not complete study
Time Frame: 12 weeks
Population: Participants that consented but did not completed 12 weeks of medication
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Number analyzed (Participants) | 16 | 16
Participants | 8 | 6

4. Secondary Outcome: Impact of Omega-3 Supplement on Post-covid Symptoms - Shortness of Breath
Description: Self-reported shortness of breath as captured at baseline (self-completing survey-pre) and after 12 weeks of treatment with omega-3 (self-completing survey-post).
Time Frame: 12 weeks from baseline
Population: Number of participants experiencing shortness of breath at 12 weeks post treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Number analyzed (Participants) | 8 | 10
Participants | 3 | 5

5. Secondary Outcome: Impact of Omega-3 Supplement on Post-covid Symptoms - Cough
Description: Self-reported cough as captured at baseline (self-completing survey-pre) and after 12 weeks of treatment with omega-3 (self-completing survey-post).
Time Frame: 12 weeks from baseline
Population: Number of participants experiencing cough at 12 weeks post treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Number analyzed (Participants) | 7 | 10
Participants | 2 | 3

6. Secondary Outcome: Impact of Omega-3 Supplement on Post-covid Symptoms - Fatigue
Description: Self-reported fatigue as captured at baseline (self-completing survey-pre) and after 12 weeks of treatment with omega-3 (self-completing survey-post).
Time Frame: 12 weeks from baseline
Population: Number of participants experiencing fatigue at 12 weeks post treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Number analyzed (Participants) | 7 | 10
Participants | 5 | 5

7. Secondary Outcome: Impact of Omega-3 Supplement on Post-covid Symptoms - Loss of Smell
Description: Self-reported loss of smell as captured at baseline (self-completing survey-pre) and after 12 weeks of treatment with omega-3 (self-completing survey-post).
Time Frame: 12 weeks from baseline
Population: Number of participants experiencing loss of smell at 12 weeks post treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Number analyzed (Participants) | 7 | 10
Participants | 4 | 3

8. Secondary Outcome: Impact of Omega-3 Supplement on Post-covid Symptoms - Loss of Taste
Description: Self-reported loss of taste as captured at baseline (self-completing survey-pre) and after 12 weeks of treatment with omega-3 (self-completing survey-post).
Time Frame: 12 weeks from baseline
Population: Number of participants experiencing loss of taste at 12 weeks post treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
Number analyzed (Participants) | 6 | 10
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: During the 12 weeks of the treatment with omega-3/placebo
Description: Self-reporting adverse events
Arm/Group | Study Arm - Omega 3 Supplement | Control Arm - Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm - Omega 3 Supplement (N=16) | Control Arm - Placebo (N=16)
Excessive Fatigue (General disorders) | 1 (1) | 0 (0)
Minimal bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (2) — Minimal gum bleeding
Bloody nose (Blood and lymphatic system disorders) | 0 (0) | 1 (4)
Localized pain (Nervous system disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT05121766/Prot_SAP_000.pdf